CLINICAL TRIAL: NCT07079592
Title: A Deep-Learning-Enabled Electrocardiogram for Detecting Pulmonary Hypertension: A Randomized Controlled Trial
Brief Title: A Deep-Learning-Enabled Electrocardiogram for Detecting Pulmonary Hypertension
Acronym: ADDPH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Pang-Yen, Liu, Assistant professor, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AI-PH
Record Dates: First submitted 2025-07-14; First posted 2025-07-23 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Artificial Intelligence (AI); Artificial Intelligence (AI) in Diagnosis; Hypertension, Pulmonary
Keywords: Artificial intelligence; electrocardiogram; deep learning; pulmonary hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Intervention Model Description: Participants undergo screening using the AI-ECG system. Those identified as high-risk for pulmonary hypertension receive echocardiography to confirm the diagnosis and guide subsequent management.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-ECG guidance (Experimental): Participants in this arm undergo screening using the AI-ECG system. Those identified as high-risk for pulmonary hypertension receive echocardiography to confirm the diagnosis and guide subsequent management.
  Interventions: Diagnostic Test: AI-ECG Guidance
- Standard clinical care (No Intervention): Participants in this arm are screened using the AI-ECG system, but diagnosis and management follow the usual clinical practice without echocardiography.

INTERVENTIONS:
Diagnostic Test: AI-ECG Guidance — Participants undergo screening using the AI-ECG system. Those identified as high-risk for pulmonary hypertension receive echocardiography to confirm the diagnosis and guide subsequent management.
  Arms: AI-ECG guidance

SUMMARY:
This study aims to validate the use of an artificial intelligence-enabled electrocardiogram (AI-ECG) to screen for elevated PAP. We hypothesize that the AI-ECG model can early identify patients with pulmonary hypertension in high-risk patients, prompting further evaluation through echocardiography, potentially resulting in improving cardiovascular outcomes.

DETAILED DESCRIPTION:
Pulmonary hypertension is often underdiagnosed due to extensive category of etiology. The diagnosis and treatment of pulmonary hypertension have changed dramatically through the re-defined diagnostic criteria and advanced drug development in the past decade. The application of Artificial Intelligence for the detection of elevated pulmonary arterial pressure (ePAP) was reported recently. An AI model based on electrocardiograms (ECG) has shown promise in not only detecting ePAP but also in predicting future risks related to cardiovascular mortality.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, ≥ 50 to 85 years of age
* At least one 12-lead ECG within 3 months

Exclusion Criteria:

* A diagnosis of PH WHO Groups 1, 2, 3, 4, or 5
* A diagnosis of hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, cardiac amyloidosis, or infiltrative cardiomyopathy
* Prior heart, lung, or heart-lung transplants
* Any systolic pulmonary artery pressure >50 mmHg by echocardiography before
* No echocardiography in 3 months before index ECG

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8666 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Pulmonary arterial pressure > 50 mmHg | 90 days
  The composite endpoint is defined as detecting pulmonary hypertension > 50mmHg by echocardiography, indicating high risk for pulmonary hypertension.

SECONDARY OUTCOMES:
Left atrial enlargement on a parasternal long axis view | Within 90 days after randomization.
  The endpoint measures the size of left atrium > 40mm on a parasternal long axis view by echocardiography.
Left atrial enlargement by left atrium volume index | Within 90 days after randomization.
  The endpoint measures the size of left atrium volume index > 29 mL/m2 in sinus rhythm or > 40 mL/m2 in AF by echocardiography.
Right ventricular enlargement on a parasternal long axis view | Within 90 days after randomization.
  The endpoint measures the size of right ventricular basal dimension > 27mm by echocardiography.
New onset of left ventricular dysfunction | Within 90 days after randomization.
  The endpoint measures the number and proportion of LVEF < 50%.

CONTACTS AND LOCATIONS:
Overall Officials: Chin Lin, associate professor, Study Director — National Defense Medical Center, Taiwan
Locations (1):
- National Defense Medical Center, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Liu PY, Hsing SC, Tsai DJ, Lin C, Lin CS, Wang CH, Fang WH. A Deep-Learning-Enabled Electrocardiogram and Chest X-Ray for Detecting Pulmonary Arterial Hypertension. J Imaging Inform Med. 2025 Apr;38(2):747-756. doi: 10.1007/s10278-024-01225-4. Epub 2024 Aug 13. PMID 39136826